CLINICAL TRIAL: NCT06108102
Title: International Post Stroke Epilepsy Research Repository to Characterize Post-stroke Epilepsy Population and Their Outcomes
Brief Title: International Post-Stroke Epilepsy Research Repository
Acronym: IPSERR
Status: Enrolling by invitation | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Monash University (Other)
Responsible Party: Sponsor
Other Study IDs: 2000032731; No NIH funding (Other: 11.15.23)
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Post Stroke Epilepsy; Post Stroke Seizure; Stroke; Epilepsy
Keywords: Post-stroke epilepsy; Clinical outcomes; Prognosis; Individual patient data
MeSH Terms: conditions — Stroke; Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-stroke epilepsy: Stroke patients aged ≥18 years, with ischemic or hemorrhagic stroke, presenting with early or late onset post-stroke seizures.
  Interventions: Other: Presence of stroke, either ischemic or hemorrhagic (intracerebral and subarachnoid)
- No post-stroke epilepsy: Stroke patients aged ≥18 years, with ischemic or hemorrhagic stroke, presenting with no post-stroke seizures.
  Interventions: Other: Presence of stroke, either ischemic or hemorrhagic (intracerebral and subarachnoid)

INTERVENTIONS:
Other: Presence of stroke, either ischemic or hemorrhagic (intracerebral and subarachnoid) — Presence of ischemic or hemorrhagic stroke confirmed by neuroimaging and clinical diagnosis

SUMMARY:
The International Post-Stroke Epilepsy Research Repository (IPSERR): The study aims to collate and categorize data reported by post-stroke epilepsy (PSE) researchers and lodge it within the IPSERR. Using the IPSERR database, we will conduct two individual patient data (IPD) analyses: (1) determine epilepsy, functional, and cognitive outcomes in stroke patients who develop post-stroke seizure and (2) build and validate post-stroke epilepsy prediction model and compare performance against existing models.

DETAILED DESCRIPTION:
The cerebrovascular disease is the most common cause of late-onset epilepsy. PSE is associated with increased morbidity, including cognitive decline, dependence, and poor quality of life, and is a critical determinant factor of stroke prognosis. We recently reported a systematic review and meta-analysis of 71 papers that suggested that post-stroke seizures are associated with more significant mortality and poor functional and cognitive outcomes (PMID:37721736). In this study, we observed disparate methods used by the individual investigators. We also noted variations in study reporting. PI aims to analyze existing individual patient data, including those analyzed in the systematic review, by collaborating with colleagues in the field and developing IPSERR into a resource for future collaborative studies that will tackle anti-epileptogenesis drug trial design.

Design and Rationale:

1. International Post-Stroke Epilepsy Research Repository (IPSERR): The PI convened the International Post-Stroke Epilepsy Research Consortium (IPSERC) with co-convenor Dr. Patrick Kwan, Monash University, Australia. IPSERR was subsequently founded to collect retrospective and prospective PSE data to promote all aspects of PSE research. Participating centers will obtain legal approvals for human subject research as per the requirements of their jurisdiction. The PI (NKM) has IRB approval for IPSERR. A data use agreement (DUA) will be executed to receive data. The PI will invite the authors of all 71 papers in the systematic review to join IPSERC and request them to contribute data to IPSERR. A protocol (including the charter) for the proposed IPD analyses has been accepted for publication and will be available to the collaborators for review.
2. The PI will use the Yale Center for Research Computing (YCRC) resources to manage IPSERR's clinical, radiological, and electrophysiological data.
3. The PI will use Redcap for clinical data management. The Redcap server is housed within the Yale-New Haven Hospital secured data center behind their firewall. The databases are encrypted at rest for HIPAA compliance. Full database backups are made twice daily, seven days a week.
4. Study duration: 2023-2029
5. Rationale: Collaboration is vital for PSE research. This is because approximately 10% of stroke patients develop PSE. Together, investigators can collect a large sample of the PSE patient population and conduct robust analyses to draw meaningful conclusions. The collation of IPD from many different sources involving different interventions and stroke subpopulations will strengthen our ability to provide data for future research on many topics relating to PSE. The availability of high-speed internet has made it easier than ever to work closely with colleagues worldwide and share data. There are many examples of such successful efforts. For example, PI Dr. Mishra closely worked with the SITS-ISTR registry at Karolinska University, Stockholm, and the Virtual Stroke Trials Archive (VISTA) at the University of Glasgow, UK. These two international efforts recorded tPA and stroke trial data, respectively, and provided them for testing several hypotheses. Dr. Mishra subsequently worked at the US FDA, where he was exposed to other large collaborative scientific efforts like MDEpiNET. The PI seeks to capitalize on his experiences, network of colleagues worldwide, and recent technological advancement in data science to build the IPSERR. We anticipate that the IPSERR will bring together large datasets from previously conducted PSE research that would otherwise ordinarily remain dormant. The PI will request data from the authors of papers included in the systematic review (N=71 papers reporting approximately 20000 PSE patient data) and from the IPSERC members. The PI will report IPSERR in the first year and the results of the two research projects anchored on it in the second year. The PI will recognize that not all authors of the previously published literature in our systematic review will have data to share. However, even if 20% of the patient data is obtained from those studies, the PI expects an extensive database of approximately 8000 patients. With this success, the PI expects the IPSERR to continue growing. IPSERR will catalytically advance PSE research because it will provide the PSE research community with an extensive database for hypotheses testing and a framework to anchor future prospective studies.

ELIGIBILITY:
Inclusion Criteria:

* Studies with minimum dataset of 100 patients
* Studies comprising stroke patients aged ≥18 years, with ischemic or hemorrhagic stroke, presenting early or late PSS with data on patient outcome measures.
* Documented consent or waiver of consent following local Institutional Review Board-approved procedure.
* Studies published on human subjects.
* No restriction based on the date or language of publication, gender, or ethnicity.

Exclusion Criteria:

* Studies of patients with a prior history of seizures before the index stroke,
* Studies that did not report outcome data, or are not able to share IPD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stroke aged ≥18 years, with ischemic or hemorrhagic stroke, presenting with early or late post-stroke seizures. Patients presenting ≤1 week will be classified as early seizures and >1 week will be classified as late seizures.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Mortality (modified Rankin Scale = 6) | At 1 year, 2 year, and 5 year follow-up
  The modified Rankin Scale (mRS) is a clinician-reported measure of global disability for evaluating recovery from stroke. It ranges from 0 (no symptoms) to 6 (death).
Poor functional outcome (modified Rankin Scale 3-6) | At 1 year, 2 year, and 5 year follow-up
  The modified Rankin Scale (mRS) is a clinician-reported measure of global disability for evaluating recovery from stroke. It ranges from 0 (no symptoms) to 6 (death), with 0-2 indicating a good functional outcome and 3-6 indicating a poor functional outcome.
Seizure frequency | At 1 year, 2 year, and 5 year follow-up
  Number of seizures post-stroke identified clinically or based on an electroencephalogram (EEG).
Seizure severity | At 1 year, 2 year, and 5 year follow-up
  Defined by impaired awareness and the presence of bilateral tonic or clonic seizures.
Occurrence or frequency of status epilepticus | At 1 year, 2 year, and 5 year follow-up
  Status epilepticus is defined as a seizure or series of seizures lasting more than 30 minutes without recovery of consciousness based on electroencephalogram (EEG) findings.
Length of hospital stay | At 1 year, 2 year, and 5 year follow-up
  The duration of hospital admission for a stroke is measured in days.
Cognitive decline assessed on an 11-question Mini-Mental State Examination (MMSE) tool or a 30-point Montreal Cognitive Assessment (MoCA) scale | At 1 year, 2 year, and 5 year follow-up
  MMSE is tests cognitive function. It is scored out of 30, with a score of ≤26 indicating cognitive impairment. MoCA assesses mild cognitive dysfunction. It is scored out of 30, with a score of ≤24 indicating cognitive impairment.

SECONDARY OUTCOMES:
Recurrent stroke | At 1 year, 2 year, and 5 year follow-up
  A diagnosis of a subsequent stroke will be made based on neuroimaging.
Antiseizure medication discontinuation | At 1 year, 2 year, and 5 year follow-up
  Switching of antiseizure medication (ASM) defined as discontinuation of one ASM and starting of another due to adverse events or treatment ineffectiveness.
Treatment adverse events | At 1 year, 2 year, and 5 year follow-up
  Adverse events are defined as any side effects occurring due to antiseizure medication administration during the course of the study.
Depression assessed on 21-item Hamilton Depression Rating Scale (HAM-D) | At 1 year, 2 year, and 5 year follow-up
  HAM-D is a tool used to assess depression symptoms. Depression post-ASM administration is defined as HAM-D score of 0-13 mild; 14-17 mild to moderate; >17 moderate to severe depression.
Anxiety assessed on 14-item Hamilton Anxiety Rating Scale (HAM-A) | At 1 year, 2 year, and 5 year follow-up
  HAM-A is a psychological questionnaire that measures the severity of a patient's anxiety. Anxiety post-ASM administration is defined as HAM-A score of <17 mild; 18-24 moderate; 25-30 moderate to severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Nishant K Mishra, MD PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided
The PI (NKM) will create a centralized database, collect, and analyze PSE patient data, and establish common data protocols. IPSERR welcomes all PSE researchers as impartial members, granting membership to institutions. Each organization will have a role in the IPSERR steering committee. One named individual, usually the principal investigator of the contributing study, will represent the institution in the IPSERR. Steering committee members will review and approve research proposals. To address data concerns like confidentiality, reliability, and authorship, strict guidelines will be set for handling patient data, promoting ethical data sharing and collaborators' involvement in publications. Data will be securely stored, and access will be restricted to authorized individuals. The IPSERR constitution will define eligibility, data protection, storage, compatibility, and documentation.

REFERENCES:
- [Background] Mishra NK, Kwan P, Tanaka T, Sunnerhagen KS, Dawson J, Zhao Y, Misra S, Wang S, Sharma VK, Mazumder R, Funaro MC, Ihara M, Nicolo JP, Liebeskind DS, Yasuda CL, Cendes F, Quinn TJ, Ge Z, Scalzo F, Zelano J, Kasner SE; International Post-Stroke Epilepsy Research Consortium (IPSERC); International Post Stroke Epilepsy Research Consortium (IPSERC). Clinical characteristics and outcomes of patients with post-stroke epilepsy: protocol for an individual patient data meta-analysis from the International Post-stroke Epilepsy Research Repository (IPSERR). BMJ Open. 2023 Nov 15;13(11):e078684. doi: 10.1136/bmjopen-2023-078684. PMID 37968000